CLINICAL TRIAL: NCT05959681
Title: Longitudinal Trial Assessing Cellulite in Women Wearing a New Compression Garment - One Side With Ink Printed Micro-pads ("Vari-pads") and One Side Without.
Brief Title: Longitudinal Trial Assessing Cellulite in Women Wearing a New Compression Garment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Whiteley Clinic (Other)
Responsible Party: Principal Investigator, Mark Whiteley, Medical Director of The Whiteley Clinic, The Whiteley Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TWC-SM-2023-01
Record Dates: First submitted 2023-06-28; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Cellulite
Keywords: compression
MeSH Terms: conditions — Cellulite

STUDY DESIGN:
Intervention Model Description: Prospective observational cohort study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Cohort (Experimental): A cohort of 60 biological females who volunteered to be part of the 6 months study.
  Interventions: Device: Compression garment with Vari-pad microdots ink-printed on inside.

INTERVENTIONS:
Device: Compression garment with Vari-pad microdots ink-printed on inside. — Initially, participants wear a garment with Vari-pads on one side (left or right) only and swap to a garment with Vari-pads on both sides if / when the participants notice a difference between the sides. Wearing garment 8 hours per 24 hours.

SUMMARY:
The investigators are investigating a compression garment that appears to reduce the appearance of Cellulite. The garment has both compression and patented ink-printed micro-dots ("Vari-pads"). These Vari-pads on the inner aspect of the garment are thought to increase the lymphatic return over compression alone.

In this study, volunteers with cellulite are asked to wear the garment, with only one side (left or right) having the active Vari-pads. The participants wear the garment for at least 8 hours per day. If, and when, the participants notice a difference between the sides (left and right sides), the participants will notify the investigators. At this point the participants will be invited to the trial centre for an assessment and to be swapped to a garment with Vari-pads on both sides.

Apart from this variable end-point, the participants will be reviewed routinely at 3 and 6 months. The trial ends at 6 months.

DETAILED DESCRIPTION:
The product being tested is to be a retail (non-medical) garment. This garment is a pair of standard compression shorts with a pattern of small, raised pads ("Vari-pads") of different heights printed on the inner aspect. A previous trial has suggested that wearing this garment for over eight hours a day can reduce the appearance of cellulite. In addition, participants found these compression pants to be very comfortable.

In this proposed trial, the investigators wish to investigate whether the previously found subjective and objective improvement of the appearance of cellulite is due to the compression alone, or whether the Vari-pads on the inside of the product enhance the subjective or objective impression of cellulite. As such, the investigators have asked the manufacturer to produce 60 pairs of pants where the Vari-pads are printed onto the inner aspects as per usual on one side, but not on the other side. On this other side, there will be a dot of the same colour printed, but it will not be raised.

The participants will be asked to wear the apparel for eight hours or more a day, at times that the participants find most suitable.

If and when the participants notice a difference in the appearance of cellulite between the right and left side, the participants will notify the investigators. At this point the investigators will invite the participants to the trial centre for an assessment. The participants will be swapped into the normal garments which have Vari-pads on both sides. The participants will then wear these garments for the remainder of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Biological females, over the age of 18 years old, who are able to walk normally and who have cellulite on their buttocks and/or upper thighs.

Due to having to produce special garments for this trial where only half of the garment has the Vari-pads, there will be for following restrictions:

Total number = 60.

Volunteers will be asked their sizes (Small, Medium, Large and Extra large) and will only be invited to attend if there are available places in that category.

Sizes:

* Small = 10
* Medium = 20
* Large = 20
* Extra large = 10

Exclusion Criteria:

* Women under 18 years of age.
* Women who are pregnant or who intend to get pregnant in the next 6 months.
* Women with no discernible cellulite on initial examination.
* Women undergoing any other treatment which aims to reduce the appearance of cellulite.
* Women who are unable to complete at least 3 months of this trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Time to subjective improvement on side with Vari-pads | 0-6 months
  Time to notice difference in cellulite between the sides when wearing garment with one side having Vari-pads.

SECONDARY OUTCOMES:
Quality of life changes | 0-6 months
  Quality of life changes by Celluqol® questionnaire at 0, 3 and 6 months.
  The Celluqol tool gives a numerical outcome 8-40:
  From 8 to 16 points - cellulite does not affect quality of life From 16 to 24 points - cellulite slightly affects quality of life From 24 to 32 points - cellulite reasonably affects quality of life From 32 to 40 points - cellulite intensely affects quality of life
Objective clinical assessement of photographs by 2 blinded observers | 0-6 months
  Changes in photographs 0,3,6 months as assessed by 2 blinded observers who are clinicans expereinced in cellulite assessment. Each photograph will be blinded by a numerical code and blinded assessment will be by scoring 0-10. 0 is the worst posisble cellulite and 10 being no cellulite visible at all.
Transcutaneous water content | 0-6 months
  Changes in transcutaneous water measurements - this is a numerical meaurement direct from the device.

CONTACTS AND LOCATIONS:
Locations (1):
- The Whiteley Clinic, Guildford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arora G, Patil A, Hooshanginezhad Z, Fritz K, Salavastru C, Kassir M, Goldman MP, Gold MH, Adatto M, Grabbe S, Goldust M. Cellulite: Presentation and management. J Cosmet Dermatol. 2022 Apr;21(4):1393-1401. doi: 10.1111/jocd.14815. Epub 2022 Feb 14. PMID 35104044
- [Background] Kiely MJ, Poulsen A, Muschamp SD, Sallis C, Whiteley MS. Participant Reported Improvement in Cellulite by Vari-Pad Apparel and Objective Measurements - A "First Use" Pilot Study. Clin Cosmet Investig Dermatol. 2023 Sep 20;16:2573-2583. doi: 10.2147/CCID.S426978. eCollection 2023. PMID 37750084
- [Background] Nurnberger F, Muller G. So-called cellulite: an invented disease. J Dermatol Surg Oncol. 1978 Mar;4(3):221-9. doi: 10.1111/j.1524-4725.1978.tb00416.x. PMID 632386
- [Background] Hexsel D, Weber MB, Taborda ML, Dal'Forno T, do Prado DZ. Celluqol® - a quality of life measurement for patients with cellulite. Surgical and Cosmetic Dermatology 2011 (Jan);3(2):96-101

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2023-06-28): https://cdn.clinicaltrials.gov/large-docs/81/NCT05959681/Prot_ICF_000.pdf